CLINICAL TRIAL: NCT04637191
Title: Cognitive Function Evaluation and Rehabilitation by a Digital Game: MentalPlus®
Acronym: MentalPlus®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: University of Copenhagen (Other); Max Planck Institute for Human Development (Other); Karolinska Institutet (Other); The Cleveland Clinic (Other); University of California, Los Angeles (Other); UMC Utrecht (Other); Harvard Medical School (HMS and HSDM) (Other); Keio University (Other); California Institute of Technology (Other)
Responsible Party: Principal Investigator, Livia Stocco Sanches Valentin, Professor, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: USaoPaulo-I
Record Dates: First submitted 2017-05-30; First posted 2020-11-19 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Neuropsychological Test
Keywords: Digital games; Neuropsychology; Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MentalPlus® (Experimental): This group performed the task in the digital game for 25 minutes and later will be evaluated with standardized and validated neuropsychological tests for the studied population.
  Interventions: Device: MentalPlus®

INTERVENTIONS:
Device: MentalPlus® — A digital game named MentalPlus will be used to evaluate the possibility of this game becoming a neuropsychological test.
  Other Names: Digital Game

SUMMARY:
Cognitive dysfunction is a frequent adverse event in the postoperative period, especially in elderly patients. The tests commonly used for the detection of postoperative cognitive dysfunction (POCD) are time-consuming, which limits routine use. Consequently, there is a limitation to adopting measures to increase preoperative cognitive reserve and rehabilitation of POCD. That situation incentivizes searching for alternative diagnosis methods to overcome that limitation. Digital games have potential neuromodulator effects and have been used as an alternative to psychotherapeutic treatment. However, the tests used to detect postoperative cognitive dysfunction (POCD) are time-consuming, making it difficult to implement routine screening measures. This presents a challenge for increasing preoperative cognitive reserve and rehabilitating POCD. Researchers are exploring alternative diagnostic methods, such as digital games, to address this challenge. Digital games have potential neuromodulator effects and are an alternative to psychotherapeutic treatments and cognitive rehabilitation. This study aims to validate MentalPlus®, a digital game, as a tool for cognitive assessment, POCD evaluation, and POCD rehabilitation-habilitation of mental skills. It is hypothesized that a digital game could replace the usual neuropsychological tests for detecting POCD.

DETAILED DESCRIPTION:
METHODS: The research subject that will be studied might present some characteristics: over 20 years old, literate, of both genders, and candidate for surgery under general anesthesia in the Hospital das Clínicas of the Faculty of Medicine, University of São Paulo. Reliability MentalPlus® analysis will be performed as the first part of the study with healthy volunteers. Later, the volunteers assess cognitive functions, like memory, attention, and executive functions, using a usual psychological test battery. Compare the psychological test battery results with MentalPlus® video game scores. The MentalPlus® digital game will be applied to all study phases. A third project will use functional magnetic resonance imaging (fMRI) to assess the association between brain response and cognitive training by MentalPlus®.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who accept the invitation will be first submitted to the TICS Instrument (Telephone Interview Cognitive Status), which aims to verify the global cognitive status of the subject evaluated. Will be included subjects with TICS score >25.

Exclusion Criteria:

* Patients who do not meet the TICS inclusion criteria will be excluded at this stage and informed that they did not fulfill all the requirements for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
Validation of MentalPlus® digital game as a neuropsychological test for assess cognitive functions: executive, attention, memory and language. | 1 year
  Cognitive evaluation of 60 patients in the pre and postoperative period using the MentalPlus scale for the evaluation of postoperative cognitive dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Livia S Valentin, Ph.D, Principal Investigator — University of Sao Paulo School of Medicine
Locations (1):
- Livia Stocco Sanches Valentin, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hudetz JA, Iqbal Z, Gandhi SD, Patterson KM, Hyde TF, Reddy DM, Hudetz AG, Warltier DC. Postoperative cognitive dysfunction in older patients with a history of alcohol abuse. Anesthesiology. 2007 Mar;106(3):423-30. doi: 10.1097/00000542-200703000-00005. PMID 17325499
- [Background] Youngblom E, DePalma G, Sands L, Leung J. The temporal relationship between early postoperative delirium and postoperative cognitive dysfunction in older patients: a prospective cohort study. Can J Anaesth. 2014 Dec;61(12):1084-92. doi: 10.1007/s12630-014-0242-6. Epub 2014 Oct 7. PMID 25287962
- [Background] Boos GL, Soares LF, Oliveira Filho GR. [Postoperative cognitive dysfunction: prevalence and associated factors.]. Rev Bras Anestesiol. 2005 Oct;55(5):517-24. doi: 10.1590/s0034-70942005000500006. Portuguese. PMID 19468642
- [Background] Burkhart CS, Steiner LA. Can postoperative cognitive dysfunction be avoided? Hosp Pract (1995). 2012 Feb;40(1):214-23. doi: 10.3810/hp.2012.02.962. PMID 22406897
- [Background] Damuleviciene G, Lesauskaite V, Macijauskiene J. [Postoperative cognitive dysfunction of older surgical patients]. Medicina (Kaunas). 2010;46(3):169-75. Lithuanian. PMID 20516755
- [Background] Blumberg FC, Fisch SM. Introduction: digital games as a context for cognitive development, learning, and developmental research. New Dir Child Adolesc Dev. 2013 Spring;2013(139):1-9. doi: 10.1002/cad.20026. PMID 23483688
- [Background] Green CS, Bavelier D. Learning, attentional control, and action video games. Curr Biol. 2012 Mar 20;22(6):R197-206. doi: 10.1016/j.cub.2012.02.012. PMID 22440805
- [Background] Fernandez-Aranda F, Jimenez-Murcia S, Santamaria JJ, Gunnard K, Soto A, Kalapanidas E, Bults RG, Davarakis C, Ganchev T, Granero R, Konstantas D, Kostoulas TP, Lam T, Lucas M, Masuet-Aumatell C, Moussa MH, Nielsen J, Penelo E. Video games as a complementary therapy tool in mental disorders: PlayMancer, a European multicentre study. J Ment Health. 2012 Aug;21(4):364-74. doi: 10.3109/09638237.2012.664302. Epub 2012 May 1. PMID 22548300
- [Background] Kuhn S, Lorenz R, Banaschewski T, Barker GJ, Buchel C, Conrod PJ, Flor H, Garavan H, Ittermann B, Loth E, Mann K, Nees F, Artiges E, Paus T, Rietschel M, Smolka MN, Strohle A, Walaszek B, Schumann G, Heinz A, Gallinat J; IMAGEN Consortium. Positive association of video game playing with left frontal cortical thickness in adolescents. PLoS One. 2014 Mar 14;9(3):e91506. doi: 10.1371/journal.pone.0091506. eCollection 2014. PMID 24633348
- [Background] Kuhn S, Gleich T, Lorenz RC, Lindenberger U, Gallinat J. Playing Super Mario induces structural brain plasticity: gray matter changes resulting from training with a commercial video game. Mol Psychiatry. 2014 Feb;19(2):265-71. doi: 10.1038/mp.2013.120. Epub 2013 Oct 29. PMID 24166407
- [Background] Saleem M, Anderson CA, Gentile DA. Effects of Prosocial, Neutral, and Violent Video Games on Children's Helpful and Hurtful Behaviors. Aggress Behav. 2012 Jul-Aug;38(4):281-7. doi: 10.1002/ab.21428. PMID 25363697
- [Background] Montag C, Weber B, Trautner P, Newport B, Markett S, Walter NT, Felten A, Reuter M. Does excessive play of violent first-person-shooter-video-games dampen brain activity in response to emotional stimuli? Biol Psychol. 2012 Jan;89(1):107-11. doi: 10.1016/j.biopsycho.2011.09.014. Epub 2011 Oct 5. PMID 21982747
- [Background] Gentile DA, Choo H, Liau A, Sim T, Li D, Fung D, Khoo A. Pathological video game use among youths: a two-year longitudinal study. Pediatrics. 2011 Feb;127(2):e319-29. doi: 10.1542/peds.2010-1353. Epub 2011 Jan 17. PMID 21242221
- [Background] Bavelier D, Green CS, Pouget A, Schrater P. Brain plasticity through the life span: learning to learn and action video games. Annu Rev Neurosci. 2012;35:391-416. doi: 10.1146/annurev-neuro-060909-152832. PMID 22715883
- [Background] Oei AC, Patterson MD. Enhancing cognition with video games: a multiple game training study. PLoS One. 2013;8(3):e58546. doi: 10.1371/journal.pone.0058546. Epub 2013 Mar 13. PMID 23516504
- [Background] Boot WR, Blakely DP, Simons DJ. Do action video games improve perception and cognition? Front Psychol. 2011 Sep 13;2:226. doi: 10.3389/fpsyg.2011.00226. eCollection 2011. PMID 21949513
- [Background] Merabet LB, Connors EC, Halko MA, Sanchez J. Teaching the blind to find their way by playing video games. PLoS One. 2012;7(9):e44958. doi: 10.1371/journal.pone.0044958. Epub 2012 Sep 19. PMID 23028703
- [Background] Thompson JJ, Blair MR, Chen L, Henrey AJ. Video game telemetry as a critical tool in the study of complex skill learning. PLoS One. 2013 Sep 18;8(9):e75129. doi: 10.1371/journal.pone.0075129. eCollection 2013. PMID 24058656
- [Background] Sanchez CA. Enhancing visuospatial performance through video game training to increase learning in visuospatial science domains. Psychon Bull Rev. 2012 Feb;19(1):58-65. doi: 10.3758/s13423-011-0177-7. PMID 22037919
- [Background] Mathewson KE, Basak C, Maclin EL, Low KA, Boot WR, Kramer AF, Fabiani M, Gratton G. Different slopes for different folks: alpha and delta EEG power predict subsequent video game learning rate and improvements in cognitive control tasks. Psychophysiology. 2012 Dec;49(12):1558-70. doi: 10.1111/j.1469-8986.2012.01474.x. Epub 2012 Oct 23. PMID 23095124
- [Background] Maclin EL, Mathewson KE, Low KA, Boot WR, Kramer AF, Fabiani M, Gratton G. Learning to multitask: effects of video game practice on electrophysiological indices of attention and resource allocation. Psychophysiology. 2011 Sep;48(9):1173-83. doi: 10.1111/j.1469-8986.2011.01189.x. Epub 2011 Mar 9. PMID 21388396
- [Background] Deveau J, Lovcik G, Seitz AR. Broad-based visual benefits from training with an integrated perceptual-learning video game. Vision Res. 2014 Jun;99:134-40. doi: 10.1016/j.visres.2013.12.015. Epub 2014 Jan 6. PMID 24406157
- [Background] Valentin LSS, Valentin TSS, Carmona MJC, Aguilar G, Pires VY, Garcia RC, et al. Digital Game Test Neuropsychology. Fundação Biblioteca Nacional. 2014.
- [Background] Valentin LSS, Valentin TSS, Carmona MJC, Garcia RC, Correa RD, Gondim GB, et al. Mental Plus. INPI - Instituto Nacional da Propriedade Intelectual. 2014.